CLINICAL TRIAL: NCT01877590
Title: Alpha-lipoic Acid Reduces Left Ventricular Mass in Normotensive Type 2 Diabetic Patients With Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Xiang Guang-da, Director of Endocrinol Dept., Wuhan General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013Wze029
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease; Left Ventricular Mass
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo group (Placebo Comparator): An identical placebo daily
- alpha-lipoic acid group (Experimental): alpha-lipoic acid 600 mg daily for one year.
  Interventions: Drug: alpha-lipoic acid

INTERVENTIONS:
Drug: alpha-lipoic acid
  Arms: alpha-lipoic acid group

SUMMARY:
Cardiovascular complications account for the highest mortality in type 2 diabetic patients, mainly due to coronary artery disease (CAD). Most of the attention in treating CAD in type 2 diabetes is understandably directed toward treating coronary artery conditions. However there are other treatable culprits in these patients.

Left ventricular hypertrophy (LVH) is widespread in type 2 diabetic patients with CAD, even in the absence of hypertension. It is a strong predictor of cardiovascular events and all-cause mortality. Regression of LVH has been associated with an improved prognosis, independent of change in blood pressure (BP). Therefore, cardiovascular events and mortality in type 2 diabetes with CAD might will be reduced if the investigators can find novel therapies to regress LVH.

Alpha-lipoic acid reduces oxidative stress which then regresses LVH. Alpha-lipoic acid can improve endothelial function in diabetic conditions. Hence, the main aim of this study was to assess whether alpha-lipoic acid could regress LVM in type 2 diabetic patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* CAD
* Left ventricular hypertrophy
* HbA1c below 7.0%
* blood pressure <130/80 mmHg

Exclusion Criteria:

* Patients were excluded if they were currently alpha-lipoic acid for one year, had a previous adverse reaction to alpha-lipoic acid.
* hey were also excluded if they had renal and liver dysfunction, heart failure, or malignancy, or were unable to give informed consent.
* Patients with contraindications to cardiac magnetic resonance (CMR) (pacemakers, claustrophobia) were also excluded, as were pregnant or lactating women.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Alpha-lipoic acid regress the left ventricular mass | one year
  Alpha-lipoic acid 600 mg daily for one year.

SECONDARY OUTCOMES:
The change of endothelial dysfunction before and after alpha-lipoic acid intervention. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan General Hospital, Wuhan, Hubei, China